CLINICAL TRIAL: NCT04145596
Title: A Phase 1 Study to Investigate a Single Bolus Dose Followed With a 30 Minute Constant Infusion of HSK3486 on the Safety and Pharmacokinetics/Pharmacodynamics of HSK3486 in Patients With Hepatic Impairment (Single-Center, Open-label, Parallel-Group)
Brief Title: Safety and Pharmacokinetics/Pharmacodynamics of HSK3486 in Patients With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Haisco Pharmaceutical Group Co., Ltd (Industry)
Collaborators: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Organization: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HSK3486-105
Record Dates: First submitted 2019-10-23; First posted 2019-10-30 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — HSK3486

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Compensated Chronic Liver Disease (Child-Pugh A) (Active Comparator)
  Interventions: Drug: HSK3486
- Decompensated Chronic Liver Disease (Child-Pugh B) (Active Comparator)
  Interventions: Drug: HSK3486
- healthy volunteers（Normal liver functions） (Active Comparator)
  Interventions: Drug: HSK3486

INTERVENTIONS:
Drug: HSK3486 — HSK3486，Initially 0.4 mg/kg was administered as a 1 minute bolus, followed immediately by a constant infusion dose of 0.4 mg/kg/h administered as a 30 minute infusion via infusion pump.

SUMMARY:
Comparison of the pharmacokinetics/Pharmacodynamics of the HSK3486 in Patients With Mild and Moderate Hepatic Impairment Compared with Healthy Volunteers

DETAILED DESCRIPTION:
This is a single-center, open-label, non-randomized, parallel-controlled Phase I clinical study carried out in patients with compensated chronic liver disease (Child-Pugh A), patients with decompensated chronic liver disease (Child-Pugh B), and age-, weight-, and gender-matched subjects with normal liver functions.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form and fully understand the content, procedure and possible adverse effects before the trial starts；
2. Able to complete the study in compliance with the requirements of the clinical trial protocol;
3. Subjects (including their partners) are willing to voluntarily adopt an effective measure of contraception starting from screening to 6 months after the last dose of the investigational drug.
4. Male or female subjects aged 18-64 years old (including 18 and 64 years old);
5. Male subjects weighing ≥ 50 kg, female subjects weighing ≥ 45 kg;Body mass index (BMI) = weight (kg)/height2 (m2); BMI of ≥ 18 and ≤ 30 kg/m2 (inclusive);
6. Blood pressure between 90-149/60-94 mmHg (inclusive); heart rate between 55-100 bpm (inclusive); body temperature between 35.9-37.6°C (inclusive); respiratory rate between 12-20 breaths per min (inclusive); SpO2 when inhaling ≥ 95%;
7. Normal physical examination results or abnormal physical examination results with no clinical significance;
8. For subjects with normal liver functions, their clinical laboratory tests (blood routine, blood biochemistry, urine routine, and coagulation function) should be normal or abnormal without clinical significance;
9. No potential difficult airway (modified Mallampati score of Grade I to II);
10. For subjects with normal liver functions, they should have no history of primary diseases in major organs, including but not limited to gastrointestinal, respiratory, renal, hepatic, neurological, hematological, , endocrine, oncological, immunological, psychiatric or cardiovascular and cerebrovascular diseases;

    Patients with Hepatic Insufficiency Must Also Meet the Following Inclusion Criteria:
11. Child-Pugh grade A or B hepatic insufficiency caused by previous primary liver diseases: including non-alcoholic steatohepatitis and viral hepatitis (hepatitis B, hepatitis C);
12. The liver function is determined by the investigators as stable within 14 days before drug administration;
13. Have not used any drug or dosing regimen within 4 weeks before screening that can stabilize the primary liver disease.

Exclusion Criteria:

1. Have not used any drug or dosing regimen within 4 weeks before screening that can stabilize the primary liver disease;
2. Patient having contraindications to deep sedation/general anesthesia or a history of past sedation/anesthesia accidents;
3. Known sensitivity to excipients in HSK3486 injectable emulsion (soybean oil, glycerin, triglyceride, egg lecithin, sodium oleate and sodium hydroxide); or with allergic constitution (including history of drug allergies and allergic diseases);
4. History of alcohol abuse (> 2 units of alcohol consumed per day: 1 unit = 285 mL of beer, or 25 mL of liquor, or 100 mL of wine) within 3 months prior to screening;
5. History of drug abuse within 3 months prior to screening, or a history of long-term use of benzodiazepines;
6. Blood/plasma donation or blood loss of ≥ 200 mL, or plasma exchange within 30 days prior to screening;
7. In receipt of prescription drugs, Chinese herbal medicines, over-the-counter drugs or food supplements (such as vitamins and calcium supplements) other than contraceptives, paracetamol, non-steroidal anti-inflammatory drugs, topical over-the-counter preparations, within 2 weeks prior to screening (patients with hepatic insufficiency can also use drugs for treating primary liver diseases);
8. Participated in other drug/medical device trials within 3 month prior to screening;
9. Patients with clinically significant abnormalities in ECG (such as tachycardia/bradycardia requiring medication, II-III degree atrioventricular block or QTcF interval ≥ 450 ms (Fridericia's correction formula), or other clinically significant abnormalities determined by the clinician);
10. Female subjects in lactation or having positive serum pregnancy test results during the screening period or the trial;
11. Positive screening result of any indicators of hepatitis B surface antigen, hepatitis C antibody or hepatitis C core antigen, HIV antibody, or syphilis antibody (hepatitis B surface antigen, hepatitis C antibody or hepatitis C core antigen may be positive for patients with hepatic insufficiency);
12. Subjects with serious or clinically significant infections (such as infections of the respiratory tract or central nervous system), trauma, or major surgery within 4 weeks prior to screening;
13. Subjects expected to have surgery or hospitalization during the trial;
14. Subjects who have consumed any beverages or foods containing alcohol (or positive alcohol breath test results), grapefruit juice or methylxanthine (such as coffee, tea, cola, chocolate, and functional drinks), participated in strenuous physical activities, and with other factors that may affect drug absorption, distribution, metabolism, and excretion within 1 day prior to dose administration;
15. Subjects with positive urine drug screening results (morphine, methamphetamine, ketamine, marijuana, ecstasy pills);
16. Subjects unsuitable for arterial blood collection, such as subjects who have positive Allen's test results;
17. Subjects who are unable to fast for 8 hrs before dose administration;
18. Subjects who have used propofol, other sedatives/anesthetics, and/or opioid analgesics or compounds containing analgesics within 72 hrs prior to dose administration;
19. Subjects judged by the investigator to be unsuitable for participating in this trial for any reason.

    The Following Exclusion Criteria are Added for Patients with Hepatic Insufficiency:
20. Clinical laboratory abnormalities with clinical significance, or other clinical findings showing the following illnesses with clinically significance, including but not limited to gastrointestinal, respiratory, renal, neural, hematological, endocrine, neoplastic, immunological, psychiatric or cardiovascular and cerebrovascular diseases other than primary liver diseases;
21. Patients with liver failure, or with cirrhotic combined with hepatic encephalopathy, hepatocellular carcinoma, and esophageal and gastric variceal bleeding and other complications considered by the investigator as unsuitable for the clinical study;
22. History of liver transplantation.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-07-13 (Actual)

PRIMARY OUTCOMES:
Peak concentration (Cmax) | -30 minutes before administration until 24 hours post administration on day 1
  Cmax（a measure of the body's exposure to HSK3486）will be compared between normal hepatic function patients and Patients with Compensated Chronic Liver Disease (Child-Pugh A) or Patients with Decompensated Chronic Liver Disease (Child-Pugh B).
Area under the concentration-time curve (AUC) | -30 minutes before administration until 24 hours post administration on day 1
  AUC（a measure of the body's exposure to HSK3486）will be compared between normal hepatic function patients and Patients with Compensated Chronic Liver Disease (Child-Pugh A) or Patients with Decompensated Chronic Liver Disease (Child-Pugh B).

SECONDARY OUTCOMES:
MOAA/S(modified observer's assessment of alert /sedation) | -5 minutes before administration until 1 hours post administration on day 1
Bispectral index(BIS) | -5 minutes before administration until 1 hours post administration on day 1
Tmax | -30 minutes before administration until 24 hours post administration on day 1
  time to peak observed
Total clearance | -30 minutes before administration until 24 hours post administration on day 1
Volume of distribution | -30 minutes before administration until 24 hours post administration on day 1
blood pressure（systolic, diastolic and mean arterial pressure） | from the screening to 3 days post-dose
  safety endpoits

CONTACTS AND LOCATIONS:
Overall Officials: Yan-hua Ding, PhD, Study Director — Phase I Clinical Trial Laboratory，The First Hospital of Jilin University
Locations (1):
- Phase I Clinical Trial Laboratory, The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Qin L, Ren L, Wan S, Liu G, Luo X, Liu Z, Li F, Yu Y, Liu J, Wei Y. Design, Synthesis, and Evaluation of Novel 2,6-Disubstituted Phenol Derivatives as General Anesthetics. J Med Chem. 2017 May 11;60(9):3606-3617. doi: 10.1021/acs.jmedchem.7b00254. Epub 2017 Apr 28. PMID 28430430
- [Derived] Hu Y, Li X, Liu J, Chen H, Zheng W, Zhang H, Wu M, Li C, Zhu X, Lou J, Yan P, Wu N, Liu X, Ma S, Wang X, Ding Y, Xuan C. Safety, pharmacokinetics and pharmacodynamics of a novel gamma-aminobutyric acid (GABA) receptor potentiator, HSK3486, in Chinese patients with hepatic impairment. Ann Med. 2022 Dec;54(1):2769-2780. doi: 10.1080/07853890.2022.2129433. PMID 36217101